CLINICAL TRIAL: NCT00914745
Title: Single Center Phase I/II, Placebo Controlled, Randomized, Double-Blind Study to Treat Recurrent Herpes Labialis by Topical Treatment With Hydroxypropyl-Beta-Cyclodextrin-Ointment (HPßCD-20% Ointment)
Brief Title: Place Controlled Study to Treat Recurrent Herpes Labialis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Devirex AG (Industry)
Responsible Party: Thomas Kuendig, University Zurich
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: ZU-HPB-001
Record Dates: First submitted 2009-06-02; First posted 2009-06-05 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2011-05

CONDITIONS: Recurrent Herpes Labialis
MeSH Terms: conditions — Herpes Labialis | interventions — Ointments

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ointment — Each time about 1.5 cm ointment have to be applied on the upper lip and 1.5 cm on the lower lip, twice daily for prophylaxis for e period of 6 month.

SUMMARY:
About 80% of the worldwide population is positive on HSV antibodies. In the United States the lifetime prevalence of recurrent herpes labialis is estimated at 20% to 40%, with approximately 100 million episodes occurring in the country every year. In Switzerland about 70% of the adult population is positive on HSV-1 and about 20% is positive on HSV-2.

The Herpes simplex virus has a lipid bilayer (virus-envelope), which causes the sensitiveness, to any kind of detergents. Within this bilayer cholesterol molecules are integrated and play a crucial role in virus entry into host cells. In vitro experiments have clearly shown that the depletion of cholesterol in HSV-envelope with 2- HPßCD has inhibited the ability of the virus to infect host cells.

The aim of this clinical trial is to reduce the number of Herpes labialis relapse and to provide patients with recurrent Herpes labialis a real benefit, concerning the simple mechanism of action and the negligible side effects. Patients having problems in swallowing the antiviral pills of standard treatment, will find with 2- HPßCD a drug, that just has to be applied on the lips, which increases patient's quality of life tremendously.

* Trial with medicinal product

ELIGIBILITY:
Inclusion criteria: Patients will be enrolled in the study if they fulfill the following inclusion criteria:

1. 18 to 50 years old,
2. Medical history of Herpes labialis with lesions on the lips or in the perioral area (<1cm from the border of the lips).
3. At least eight recurrences of labial herpes during the previous year before being en-rolled in the study.
4. Ability and willingness to participate in the study.
5. Voluntary written informed consent.

Exclusion criteria: Patients who fulfill any one of the following exclusion criteria may not be enrolled in the study:

1. Females with child bearing potential who are not using a reliable, medically accepted method of birth control (e.g. surgical, intrauterine contraceptive device, birth control pill, double barrier, hormone delivery systems such as implants or injectables, condoms or diaphragm (each in combination with contraceptive creams, foams, etc.).
2. Pregnant or breast feeding female, or women planning to become pregnant during the trial.
3. Medical history of immunosuppression by radiotherapy, chemo therapy, immunomodulatory drugs, or HIV.
4. Participation in another clinical study within 30 days prior to application of 2-HPßCD.
5. Medical history of any severe diseases like hepatitis, renal or liver dysfunction, cardiovascular, gastrointestinal, malignant tumor(s), or psychiatric disorders etc., which might influence the assessments or conduct of the trial by the discretion of the investigator.
6. Intake or application of antivirals or other prohibited concomitant medication within 30 days prior to application of 2-HPßCD, or plan to take such drugs during the trial.
7. Use of anti-inflammatory medications and steroids during the course of the study.
8. Eczema herpeticatum or any history of other skin disease that would predispose to ec-zema herpeticatum.
9. Any abnormal perioral skin condition.
10. Known or suspected allergic or adverse response to the investigational product (2- HPßCD) or its excipients (PEG 400, and PEG 8000).
11. Inability to follow the study protocol.
12. Medical history of alcohol and/ or drug abuse within the previous 12 months before enrollment in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2009-04; Primary Completion 2010-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Reducing the number of Herpes labialis relapse. | June 2009 - Mai 2010

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Zurich, Switzerland